CLINICAL TRIAL: NCT02113228
Title: Assessment of Energy Metabolism in Patients With Short Bowel Syndrome Using the Doubly Labeled Water Method
Brief Title: Energy Metabolism in Patients With Short Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Julio Sergio Marchini, Full Professor of Internal Medicine Department at Ribeirão Preto Medical School, University of Sao Paulo
Other Study IDs: Process HCRP: 1822/2013; CAAE: 12271713.3.0000.5440 (Registry Identifier: Sistema Nacional de Informações sobre Ética em Pesquisa)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Short Bowel Syndrome
Keywords: Energy metabolism; Stable isotopes; Short bowel syndrome; Doubly labeled water
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Short Bowel Syndrome: Verify the total energy expenditure in patients with short bowel syndrome using the doubly labeled water method.
- Control Group: Verify the total energy expenditure in patients without short bowel syndrome using the doubly labeled water method.

SUMMARY:
This study proposes to verify the total energy expenditure in patients with short bowel syndrome using the doubly labeled water method, as well as determining the rate of oxidation of nutrients, aiming to assist the management of nutritional therapy for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Short bowel syndrome: short bowel syndrome patients with gastrointestinal transit time less or equal 30 minutes.
* Control group: patients with the same gender, presenting age and chronic diseases similar with volunteers from the group with short bowel syndrome.

Exclusion Criteria:

- Short bowel syndrome: time of bowel resection surgery less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The recruitment of volunteers with short bowel syndrome (SIC) will be done in the Hospital das Clinicas, Faculty of Medicine of Ribeirão Preto, University of São Paulo (HCFMRP / USP). These individuals will be paired with volunteers without short bowel syndrome, which will be selected at the clinics of the Hospital of the Faculty of Medicine of Ribeirão Preto, and will constitute the control group.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Assessment of total energy expenditure using the doubly labeled water method | 14 days
  After the determination of resting energy expenditure (REE), each volunteer will receive a dose of doubly labeled water (2H2 18O). A basal urine sample is collected before the intake dose and samples taken on days 1, 2, 3, 7, 12, 13, 14, thereafter. Urine samples will be analyzed by mass spectrometry (Hydra System, HIP 20-20, Europa Scientific, Cheshire, UK) in the Mass Spectrometry Laboratory of the Faculty of Medicine of Ribeirão Preto.

SECONDARY OUTCOMES:
Resting energy expenditure (REE) and body composition measurements by indirect calorimetry and electrical bioimpedance, respectively. | After 12 hours of overnight fasting
  This study also aims to measure the REE by indirect calorimetry with a Quark (Cosmed, Italy) calorimeter and the body composition by Byodinamics 450 (Biodynamics Corp., United States).
Physical activity assessment | 14 days
  An activity monitor (activPAL ®, Glasgow, UK) is used to determine physical activity. By registering the intensity and duration of each category of activities, the system adds the energy estimated to generate a value that reflects the total energy expenditure.

CONTACTS AND LOCATIONS:
Overall Officials: Julio S Marchini, PhD, Principal Investigator — Ribeirão Preto Medical School. São Paulo University (USP)
Locations (1):
- Clinical Hospital of Ribeirao Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Schoeller DA, Taylor PB, Shay K. Analytic requirements for the doubly labeled water method. Obes Res. 1995 Mar;3 Suppl 1:15-20. doi: 10.1002/j.1550-8528.1995.tb00003.x. PMID 7736285
- [Background] Frayn KN. Calculation of substrate oxidation rates in vivo from gaseous exchange. J Appl Physiol Respir Environ Exerc Physiol. 1983 Aug;55(2):628-34. doi: 10.1152/jappl.1983.55.2.628. PMID 6618956
- [Background] Ferreira IM, Braga CB, Dewulf Nde L, Marchini JS, da Cunha SF. Vitamin serum level variations between cycles of intermittent parenteral nutrition in adult patients with short bowel syndrome. JPEN J Parenter Enteral Nutr. 2013 Jan;37(1):75-80. doi: 10.1177/0148607112441800. Epub 2012 Mar 27. PMID 22457422
- [Background] Thomson AB, Chopra A, Clandinin MT, Freeman H. Recent advances in small bowel diseases: Part II. World J Gastroenterol. 2012 Jul 14;18(26):3353-74. doi: 10.3748/wjg.v18.i26.3353. PMID 22807605
- [Background] DiBaise JK, Young RJ, Vanderhoof JA. Intestinal rehabilitation and the short bowel syndrome: part 2. Am J Gastroenterol. 2004 Sep;99(9):1823-32. doi: 10.1111/j.1572-0241.2004.40836.x. PMID 15330926
- [Background] Araujo EC, Suen VM, Marchini JS, Vannucchi H. Ideal weight better predicts resting energy expenditure than does actual weight in patients with short bowel syndrome. Nutrition. 2007 Nov-Dec;23(11-12):778-81. doi: 10.1016/j.nut.2007.07.007. Epub 2007 Sep 17. PMID 17869483
- [Background] Donohoe CL, Reynolds JV. Short bowel syndrome. Surgeon. 2010 Oct;8(5):270-9. doi: 10.1016/j.surge.2010.06.004. PMID 20709285
- [Background] Ferriolli E, Pfrimer K, Moriguti JC, Lima NK, Moriguti EK, Formighieri PF, Scagliusi FB, Marchini JS. Under-reporting of food intake is frequent among Brazilian free-living older persons: a doubly labelled water study. Rapid Commun Mass Spectrom. 2010 Mar 15;24(5):506-10. doi: 10.1002/rcm.4333. PMID 20112270
- [Background] Jeppesen PB, Mortensen PB. Intestinal failure defined by measurements of intestinal energy and wet weight absorption. Gut. 2000 May;46(5):701-6. doi: 10.1136/gut.46.5.701. PMID 10764715
- [Background] Schoeller DA. Measurement of energy expenditure in free-living humans by using doubly labeled water. J Nutr. 1988 Nov;118(11):1278-89. doi: 10.1093/jn/118.11.1278. PMID 3142975
- [Background] Thompson JS, Rochling FA, Weseman RA, Mercer DF. Current management of short bowel syndrome. Curr Probl Surg. 2012 Feb;49(2):52-115. doi: 10.1067/j.cpsurg.2011.10.002. No abstract available. PMID 22244264
- [Derived] Fassini PG, Das SK, Pfrimer K, Suen VMM, Sergio Marchini J, Ferriolli E. Energy intake in short bowel syndrome: assessment by 24-h dietary recalls compared with the doubly labelled water method. Br J Nutr. 2018 Jan;119(2):196-201. doi: 10.1017/S0007114517003373. Epub 2017 Dec 22. PMID 29268807
- [Derived] Fassini PG, Nicoletti CF, Pfrimer K, Nonino CB, Marchini JS, Ferriolli E. Bioelectrical impedance vector analysis as a useful predictor of nutritional status in patients with short bowel syndrome. Clin Nutr. 2017 Aug;36(4):1117-1121. doi: 10.1016/j.clnu.2016.07.011. Epub 2016 Jul 27. PMID 27491548
- [Derived] Fassini PG, Pfrimer K, Ferriolli E, Suen VM, Marchini JS, Das SK. Assessment of energy requirements in patients with short bowel syndrome by using the doubly labeled water method. Am J Clin Nutr. 2016 Jan;103(1):77-82. doi: 10.3945/ajcn.115.122408. Epub 2015 Dec 16. PMID 26675764